CLINICAL TRIAL: NCT06489288
Title: The Safety and Efficacy of ERAS Clinical Pathway Intotally Laparoscopic Total Gastrectomy: a Multicenter, Prospective Randomized Controlled Study
Brief Title: ERAS in Totally Laparoscopic Total Gastrectomy for Gastric Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: First Hospital of China Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Peking University Cancer Hospital & Institute (Other); Tongji Hospital (Other); General Hospital of Ningxia Medical University (Other); Second Affiliated Hospital of Suzhou University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Nanfang Hospital, Southern Medical University (Other); Gansu Provincial Hospital (Other); Fudan University (Other); Changzhi People's Hospital (Other); Zhejiang University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The Second Affiliated Hospital of Shandong First Medical University (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CLASS12
Record Dates: First submitted 2024-06-11; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer; ERAS; Laparoscopic Gastrectomy
Keywords: Gastric Cancer; ERAS; Totally laparoscopic total gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Experimental): It is necessary to remove the urinary catheter before the patient awakens from anesthesia, drink water orally in the early postoperative period, and remove the drainage tube and nutrition tube in the early postoperative period
  Interventions: Other: ERAS protocol
- control group (Other): According to conventional treatment measures, there is no need for Enhanced Recovery After Surgery
  Interventions: Other: ERAS protocol

INTERVENTIONS:
Other: ERAS protocol — The ERAS process mainly includes removing the urethral catheter before the recovery of anesthesia, removing the abdominal drainage tube within 3 days after surgery, removing the nasogastric feeding tu

SUMMARY:
The number of totally laparoscopic total gastrectomy is gradually increasing, but the safety of ERAS in these term is still unknown and further multicenter randomized controlled studies are needed.

DETAILED DESCRIPTION:
The application of ERAS during the perioperative of gastric cancer surgery can reduce hospitalization time, costs, and surgical stress response without increasing complications and readmission rates, and may even have a certain effect on improving long-term survival rates of patients. However, some studies have also shown that ERAS may increase the number of postoperative readmissions while reducing hospitalization time, costs, and recovery time after surgery. At the same time, there is still no consensus on the application standards of ERAS during the perioperative period of gastric cancer surgery , and the comprehensive implementation of ERAS programs in clinical practice still faces huge challenges. With the widespread development of totally laparoscopic total gastrectomy , the advantages of laparoscopy have been recognized. Multiple center studies have confirmed the safety of ERAS programs in totally laparoscopic distal radical gastrectomy. However, due to the complexity of totally laparoscopic total gastrectomy, there is currently no multi-center study to confirm the safety of ERAS in it. In order to better apply ERAS in clinical practice, better serve patients undergoing gastric cancer surgery, and provide more centers with practical experience in ERAS and even provide evidence for the establishment of a consensus on ERAS during the perioperative of gastric cancer surgery, our center will rely on platform advantages and previous work experience and collaborate with the CLASS Research Center to conduct a prospective, multi-center clinical study to explore the safety and effectiveness of ERAS clinical pathway in patients undergoing totally laparoscopic total gastrectomy, providing a theoretical basis for further standardizing and promoting the application of ERAS concept in the perioperative clinical practice of gastric cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years;
2. ASA I-III;
3. ECOG ≤2;
4. NRS2002: 0-2;
5. Preoperative gastroscopy and pathological biopsy confirmed adenocarcinoma;
6. The clinical stage of abdominal hypotonic enhanced CT or ultrasonic gastroscopy is cT2-3N0-3M0 or cT1N+M0 or cT4aN0M0 (according to the AJCC-8thTNM tumor staging);
7. Proposed D2 total laparoscopic radical gastrectomy (without limitation on the anastomotic method);
8. All patients did not receive adjuvant radiotherapy, chemotherapy, or other cytotoxic treatments before surgery;
9. Borrmann I-III ;
10. No history of upper abdominal surgery (except for laparoscopic cholecystectomy); no history of peritonitis or pancreatitis
11. hemoglobin ≥80g/L; absolute neutrophil count (ANC) ≥1.5×109/L; platelet ≥100×109/L; ALT, AST≤1 times the upper limit of normal; ALP≤1 times the upper limit of normal; total serum bilirubin <1.5 times the upper limit of normal; serum creatinine <1 times the upper limit of normal; serum albumin ≥35g/L;

Exclusion Criteria:

1. tumors at the esophagogastric junction or gastric tumors that have invaded the pyloric canal;
2. Those with uncontrolled epilepsy, central nervous system diseases, or a history of mental disorders;
3. Severe (i.e., active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more severe congestive heart failure, or severe drug-dependent arrhythmia, or a history of myocardial infarction within the last 6 months;
4. Patients with urinary dysfunction who require long-term indwelling catheters after surgery;
5. Patients who need immunosuppressive therapy for organ transplantation;
6. Patients with severe uncontrolled recurrent infections or other severe uncontrolled concomitant diseases;
7. Moderate or severe renal impairment [creatinine clearance equal to or lower than 50ml/min (calculated according to the Cockroft and Gault equation), or serum creatinine > upper limit of normal (ULN);
8. Emergency surgery due to tumor emergencies (bleeding, perforation, obstruction);
9. Pregnant or breastfeeding women;
10. Previously diagnosed other tumors (excluding cervical cancer and cutaneous melanoma)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2656 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
QLQ-STO22 | Changes in quality of life in QLQ-STO22 before surgery, on the 7th day after surgery, and 1 ,6,12month after surgery
  Changes in quality of life in QLQ-STO22 before surgery, on the 7th day after surgery, and 1 ,6,12month after surgery
QLQ-C30 (V3.0) | Changes in quality of life in QLQ-C30 (V3.0) before surgery, on the 7th day after surgery, and 1 ,6,12month after surgery
  Changes in quality of life in QLQ-C30 (V3.0) before surgery, on the 7th day after surgery, and 1 ,6,12month after surgery
Complication rate | 1month
  Complications rate and Clavien-Dindo classification within 1 month after surgery
DFS | 1 and 3 years
  Disease-free survival rate at 1 and 3 years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No